CLINICAL TRIAL: NCT04709614
Title: Influence of Immunological and Psychological Factors on Perceived Severity of Seasonal Allergic Rhinitis Caused by Grass Pollen
Brief Title: Psychological Factors That Influence Severity of Allergic Rhinitis
Status: Completed | Type: Observational
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Sponsor
Other Study IDs: Psycho-Grass
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: skin prick test; specific IgE; patient reported outcome; psychological factor
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective biomarker of allergic rhinitis severity is necessary for monitoring disease severity and response to treatment in clinical setting and for research. We believe that psychological factors are the missing link between patient-perceived severity of allergic rhinitis and objective biomarkers. In our pilot study, several psychological factors were studied in relation to patient reported outcomes for severity of allergic rhinitis.

DETAILED DESCRIPTION:
Monitoring allergic rhinitis (AR) severity with objective biomarkers is important for the clinical management of patients as well as for research purposes. The most commonly used tool for the assessment of AR severity is the Total Nasal Symptom Score (TNSS). Objective biomarkers like skin prick test size or specific IgE levels don't correlate with TNSS.

We studied skin prick test size and specific IgE and several patient reported outcomes including symptom score, medication scores, combined score and Juniper mini rhinitis quality of life questionnaire (RQLQ). Psychometric evaluation was performed using 5 different psychological questionnaires that measure 13 different psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* positive grass pollen skin prick test (SPT) with a wheal diameter >3mm and a history of allergic rhinitis during the grass pollen seasons

Exclusion Criteria:

* positive skin prick test for perennial allergens and allergens with potentially overlapping seasons including cypress, ash/olive, plane, and nettle families

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were selected from 185 patients managed in our outpatient clinics with a presumptive diagnosis of allergic rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Symptom score | 2 months
  Symptom severity was graded on a visual analogue scale (VAS), ranging from 0 (no symptoms) to 10 (very severe symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Zidarn, MD PhD, Principal Investigator — Klinika Golnik

IPD SHARING:
Plan to Share IPD: No